CLINICAL TRIAL: NCT06835296
Title: A Phase I, Randomized, Placebo-Controlled, Sequential Single and Multiple Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral YUQ-A1007 in Healthy Volunteers
Brief Title: A Study of Oral YUQ-A1007 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allianthera (Suzhou) Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATB102
Record Dates: First submitted 2024-12-23; First posted 2025-02-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: Phase I; Randomized; Placebo-Controlled; Sequential Escalation; Safety; Tolerability; Pharmacokinetics; YUQ-A1007; Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAD (Experimental): Single Ascending Dose Stage in Healthy Volunteers， 4 cohorts will be included
  Interventions: Drug: YUQ-A1007 is a novel gut-enriched AhR agonist. This compound is undergoing preclinical development, and comprehensive nonclinical studies.
- MAD (Experimental): Multiple Ascending Dose Stage in Healthy Volunteers, two dose levels will be included
  Interventions: Drug: YUQ-A1007 is a novel gut-enriched AhR agonist. This compound is undergoing preclinical development, and comprehensive nonclinical studies.

INTERVENTIONS:
Drug: YUQ-A1007 is a novel gut-enriched AhR agonist. This compound is undergoing preclinical development, and comprehensive nonclinical studies. — Dose: Ascending doses (SAD stage: 200, 800, 1600, or 3200 mg; MAD stage: two dosages will be determined based on the results from the SAD stage) Mode of administration: Oral, once daily.

SUMMARY:
YUQ-A1007 is a novel gut-enriched AhR agonist. The nonclinical pharmacology study indicated that YUQ-A1007 has the potential to treat IBD.

YUQ-A1007 has not been evaluated in human clinical studies. This study is first-in-human (FIH) study of YUQ-A1007. The goal of this trial is to evaluate the safety, tolerability, and pharmacokinetics of oral YUQ-A1007.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to the conduct of any study-related assessments.
2. Aged 18 to 65 years, inclusive, at the time of signing the informed consent form (ICF).
3. Male and Female participants.
4. Has body mass index (BMI) as 18.5-27.9 kg/m2 with total body weight ≥ 50 kg for male participants and ≥ 45 kg for female participants at screening.
5. With normal liver and kidney functions.
6. With normal results of clinical laboratory tests or abnormal results of clinical laboratory tests deemed not clinically significant as per investigator judgement at screening and on admission to the CRU.
7. Willing and able to comply with the study requirements, including remaining at the CRU for the in-house portion of study participation.
8. Agrees not to smoke, vape, or consume tobacco or other nicotine-containing products, not to consume alcohol, not to consume beverages containing caffeine or other xanthines.
9. Is in good health based on the medical history, physical examination, vital signs measurements, laboratory tests, and 12-lead ECGs performed at screening.

Exclusion Criteria:

1. Any condition that places the participant at significantly increased risk or may compromise the study objectives.
2. Is mentally or legally incapacitated at screening.
3. History of malignant neoplasms or carcinoma in situ.
4. Has a current or chronic history of liver disease or known hepatic or biliary abnormalities.
5. Has had symptomatic herpes zoster.
6. Has a history of any known relevant allergy/hypersensitivity or intolerance.
7. Has clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions.
8. Has a sensitivity to heparin or history of heparin-induced thrombocytopenia.
9. Has a clinically significant infection.
10. Any history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological.
11. Has a clinically significant medical condition that, in the investigator's opinion, would preclude participation in the study.
12. Any clinically significant abnormality identified in the physical examination (including vital signs) or electrocardiographic testing.
13. Has a positive test for the presence of human immunodeficiency virus (HIV), hepatitis C antibody, hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to the first dose of investigational product.
14. Has active or latent tuberculosis (TB), regardless of treatment history, or positive diagnostic TB test at screening.
15. Has received treatment with a live, attenuated vaccine within 4 weeks prior to the first dose of investigational product or anticipation of need for such a vaccine during study participation.
16. Has a contraindication to blood sampling or is considered to have insufficient peripheral venous access.
17. Has donated or lost blood or blood products in volumes of 450 mL or more within 30 days.
18. Has had prior exposure to YUQ-A1007.
19. Has participated in a study of any investigational drug, device, biologic, or other agent within 30 days or 5 half-lives prior to screening, whichever is longer.
20. Has received any prescription medications, over-the-counter medications, herbal supplements, or vitamins within 30 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product.
21. Is an employee or has a family member who is an employee of the CRU and is involved in the conduct of the study and/or supervised by the investigator; or is an employee or has a family member who is an employee of the sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of YUQ-A1007 administered orally | during the intervention (about 6 months)
  Number of participants with Treatment-emergent adverse events (TEAEs), with clinically significant changes from baseline in vital signs (body temperature, blood pressure, heart rate, and respiratory rate), physical examination findings, and 12-lead electrocardiogram (ECG) parameters, and with clinically significant changes from baseline in safety laboratory assessments (hematology, clinical chemistry, urinalysis, and stool routine test)

CONTACTS AND LOCATIONS:
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No